CLINICAL TRIAL: NCT06397417
Title: Prognosis of Refractory Out-of-hospital Cardiac Arrests Treated With Extracorporeal Cardiopulmonary Resuscitation (ECMO) by the Urgent Medical Aid Service (SAMU) of Paris
Brief Title: Refractory Cardiac Arrest Treated On Field By ECMO
Acronym: ReCATOBE
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231680
Record Dates: First submitted 2024-03-28; First posted 2024-05-02 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Out-of-Hospital Cardiac Arrest; Extracorporeal Cardiopulmonary Resuscitation
Keywords: Out-of-Hospital Cardiac Arrest; Extracorporeal Cardiopulmonary Resuscitation
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: All patients over 18 years of age who will benefit from an installation or an attempt at an ECMO installation following a non-traumatic refractory cardiac arrest care by the ECMO TEAM of the Paris SAMU over a period of 20 years old. Patients' medical data will be collected for one year after their care.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — The data from hospital treatment will be used for research as well as subsequently, that is to say after discharge from the intensive care units, medical reports and correspondence with the attending physician will be used for the study.

SUMMARY:
Out-of-hospital cardiac arrest without resumption of spontaneous circulatory activity despite advanced medical resuscitation is considered refractory. Under certain well-defined conditions, today in many cities around the world and particularly in Paris, it benefits from resuscitation called ECPR (extracorporeal cardiopulmonary resuscitation). This technique consists of the installation of an extracorporeal membrane oxygenation (ECMO) device allowing organ perfusion while waiting for a resumption of cardiac activity. Since 2011, the Paris SAMU (SAMU 75) has set up a team capable of implementing ECPR for refractory out-of-hospital cardiac arrests. This team based within the SAMU of Paris at the Necker hospital (ECMO team) composed of an emergency doctor or anesthesiologist-resuscitator, a nurse anesthetist and an ambulance driver intervenes in Paris and its nearby region at the request of medical regulation. Given the growing development of this activity, it is essential to measure its effectiveness in real-life conditions.

DETAILED DESCRIPTION:
Out-of-hospital cardiac arrest without resumption of spontaneous circulatory activity despite advanced medical resuscitation is considered refractory. Under certain well-defined conditions, today in many cities around the world and particularly in Paris, it benefits from resuscitation called ECPR (extracorporeal cardiopulmonary resuscitation). This technique consists of the installation of an extracorporeal membrane oxygenation (ECMO) device allowing organ perfusion while waiting for a resumption of cardiac activity. Since 2011, the Paris SAMU (SAMU 75) has set up a team capable of implementing ECPR for refractory out-of-hospital cardiac arrests. This team based within the SAMU of Paris at the Necker hospital (ECMO team) composed of an emergency doctor or anesthesiologist-resuscitator, a nurse anesthetist and an ambulance driver intervenes in Paris and its nearby region at the request of medical regulation. Given the growing development of this activity, it is essential to measure its effectiveness in real-life conditions.

The study consists of establishing a prospective register over a period of 20 years of patients aged over 18 years, victims of refractory non-traumatic out-of-hospital cardiac arrest in the coverage area of the ECMO TEAM of the Paris SAMU.

The 1-year survival rate of patients will be measured, the functional prognosis will be evaluated and a search for associated factors will be carried out. Patients' long-term cardiac function will be collected as well as the incidence of ECPR-related complications.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have benefited from an installation or attempted installation of an extracorporeal membrane oxygenation (ECMO) device following a non-traumatic refractory cardiac arrest as part of the ECMO TEAM of the Samu de Paris during the time of the study.
* Obtaining non-opposition from the patient or a relative in the event of the patient's death or a lasting state of health preventing them from becoming aware of the study.

Exclusion Criteria:

- Minor patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who have benefited from an installation or attempted installation of an extracorporeal membrane oxygenation (ECMO) device following a non-traumatic refractory cardiac arrest as part of the ECMO TEAM of the Samu de Paris during the time of the study.
Sampling Method: Non-Probability Sample
Enrollment: 840 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2046-03 (Estimated); Study Completion 2046-03 (Estimated)

PRIMARY OUTCOMES:
Survival | 1 year
  Survival rate at 1 year after an extracorporeal cardiopulmonary resuscitation by the ECMO TEAM of the Paris SAMU.

SECONDARY OUTCOMES:
Neurological prognosis | 1 year
  Evaluation of the functional prognosis at 1 year by the score at the Cerebral Performance Category Scale. A favorable outcome is defined by a score of 1 or 2. The score on the brain performance category scale will be determined based on hospital records and/or telephone interview with the general practitioner. The CPC score: [5: death, 4: persistent vegetative state, 3: severe disability, 2: moderate disability, 1: low disability].
Quality of life assessment | 1 year
  Evaluation of the functional prognosis at 1 year by measure of the quality of life assessed by the Short Form (36) Health Survey (SF36). The SF-36 test is a standardized questionnaire for measuring quality of life. It is carried out during a follow-up medical consultation. Description of the overall SF36 score and each of its eight sections (vitality, physical functioning, bodily pain, general health perception, physical role functioning, emotional role functioning, social role functioning, mental health).
Incidence of ECPR-related complications | 1 year
  Measurement of the incidence of complications linked to ECPR (extracorporeal cardiopulmonary resuscitation) : bleeding at the cannula puncture site, lower limb ischemia, post-load pulmonary edema, bacteremia, insertion site infection.
Left ventricular ejection fraction (LVEF) | 1 year
  Assessment of long-term cardiac function based on the data from the imaging reports carried out by the downstream services and/or the telephone interview with the general practitioner or specialist doctor.
Occurrence of major cardioavscular events | 1 year
  Report of occurrence of major cardioavscular events through analysis of medical reports within one year after cardiac arrest. Major cardioavscular events are defined as : recurrence of cardiac arrest, acute coronary syndrome, ventricular rythm disorders, acute heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Herlé Raphalen, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No